CLINICAL TRIAL: NCT04809467
Title: A Phase 1b/2a Basket Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Combination Therapy With the Anti CD19 Monoclonal Antibody Tafasitamab and the PI3Kδ Inhibitor Parsaclisib in Adult Participants With Relapsed/Refractory Non Hodgkin Lymphoma or Chronic Lymphocytic Leukemia
Brief Title: A Study Evaluating Safety, PK, and Efficacy of Tafasitamab and Parsaclisib in Participants With Relapsed/Refractory Non Hodgkin Lymphoma (R/R NHL) or Chronic Lymphocytic Leukemia (CLL)
Acronym: topMIND
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A business decision was made to discontinue further enrollment. There were no safety concerns that contributed to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCMOR 0208-101; 2020-005591-35 (EudraCT Number)
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia; Non Hodgkin Lymphoma
Keywords: Relapsed or Refractory; Leukemia; tafasitamab; parsaclisib; MOR00208; INCMOR00208
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Recurrence; Leukemia | interventions — tafasitamab; parsaclisib

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tafasitamab + parsaclisib (Experimental): Participants will be assigned to disease specific cohorts based on the histology of their underlying disease.
  Cohort 1: R/R DLBCL Cohort 2: R/R MCL Cohort 3: R/R FL Cohort 4: R/R MZL Cohort 5: R/R CLL/SLL
  Interventions: Drug: tafasitamab; Drug: parsaclisib

INTERVENTIONS:
Drug: tafasitamab — tafasitamab will be administered at a protocol defined dose once a week for cycles 1-3 and every other week from cycle 4 until progression.
  Other Names: INCMOR00208
Drug: parsaclisib — parsaclisib will be administered at protocol defined dose for cycles 1 through disease progression.
  Other Names: INCB050465

SUMMARY:
The purpose of this single-arm, open-label, Phase 1b/2a, multicenter basket study is to evaluate whether tafasitamab and parsaclisib can be safely combined at the recommended Phase 2 dose (RP2D) and dosing regimen that was established for each of the 2 compounds as a treatment option for adult participants with R/R B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed R/R B-cell malignancy: DLBCL (THRLBCL, EBV-positive DLBCL of the elderly, Grade 3b FL, HGBL with MYC and BCL2 and/or BCL6 rearrangements, transformed lymphoma); MCL ((with cyclin D1 overexpression or t(11;14); FL (Grade 1, 2, 3a); MZL (extranodal, nodal, splenic) ; CLL, or SLL
* Willingness to undergo biopsy
* At least 2 prior systemic treatment regimens, including prior treatment with an anti-CD20 antibody (all cohorts) or prior treatment with a BTK inhibitor (CLL/SLL)
* Relapsed, progressive, or refractory NHL or CLL
* For NHL/SLL: Radiographically measurable nodal or extranodal disease (all cohorts except CLL)
* ECOG-PS 0 - 2
* LVEF ≥ 50%
* Adequate renal, hepatic, bone marrow function

Exclusion Criteria:

* Any other histological type of lymphoma
* Primary or secondary CNS lymphoma
* Anticancer and/or investigational therapy within the past 30 days or 5 half-lives
* Allogeneic stem cell transplantation within the past 6 months, or ASCT within 3 months before C1D1
* Previous treatment with CD19-targeted therapy or PI3K inhibitors
* Clinically significant cardiac disease
* Other malignancy within the past 3 years
* Active graft-versus-host disease
* Stroke or intracranial hemorrhage within the past 6 months
* Chronic or current active infectious disease
* Positive virus serology for HCV, HBV, HIV
* Currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Manzke, MD, Study Director — Incyte Corporation
Locations (50):
- United States (10):
  - University of Alabama At Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - Community Health Network, Inc., Indianapolis, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Cancer Center For Blood Disorders, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Alliance, New Hyde Park, New York
  - Ohio State University, Columbus, Ohio
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
- Austria (3):
  - Ordensklinikum Linz Gmbh Elisabethinen, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - Hanusch-Krankenhaus Der Wiener Gebietskrankenkasse, Vienna
- Belgium (6):
  - Institut Jules Bordet, Brussels
  - Grand Hospital de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Az Groeninge Campus Kennedylaan, Kortrijk
  - Universitair Ziekenhuis (Uz) Leuven, Leuven
  - AZ DELTA, Roeselare
- France (4):
  - University Hospital Brest, Brest
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Justus-Liebig University, Giessen
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - University Hospital Wurzburg, Würzburg
- Italy (9):
  - S Orsolas University Hospital Seragnoli Institute of Hematology, Bologna
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori, Meldola
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Naples
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale Santa Maria Delle Croci, Ravenna
  - Irccs Istituto Clinico Humanitas, Rozzano
- Spain (14):
  - Hospital General Unviersitario de Alicante, Alicante
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hopital Sant Pau, Barcelona
  - Ico Institut Catala D Oncologia, Barcelona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal (Ciocc), Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled across 16 sites in Austria, Belgium, Spain, France, and Italy. Enrollment was not fully completed due to a strategic decision by the sponsor to discontinue further enrollment in the study based on the changing treatment landscape with respect to the use of PI3Kδ inhibitors (including but not limited to parsaclisib) for treatment of NHL. Therefore the expansion phase was not opened.
Groups:
- Cohort 1: R/R DLBCL: Participants with relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL) received tafasitamab administered at 12 milligrams per kilograms (mg/kg) intravenously (IV) on Days 1, 8, 15, and 22 of Cycles 1 through 3 and then Days 1 and 15 of each 28-day cycle from Cycle 4 onward. Participants also self-administered parsaclisib at a dose of 20 mg once daily (QD) for 8 weeks, followed by a dose of 2.5 mg QD thereafter. Study treatment was administered until progression of disease, withdrawal of consent, or unacceptable toxicity.
- Cohort 2: R/R MCL: Participants with R/R mantle cell lymphoma (MCL) received tafasitamab administered at 12 mg/kg IV on Days 1, 8, 15, and 22 of Cycles 1 through 3 and then Days 1 and 15 of each 28-day cycle from Cycle 4 onward. Participants also self-administered parsaclisib at a dose of 20 mg QD for 8 weeks, followed by a dose of 2.5 mg QD thereafter. Study treatment was administered until progression of disease, withdrawal of consent, or unacceptable toxicity.
- Cohort 3: R/R FL: Participants with R/R follicular lymphoma (FL) received tafasitamab administered at 12 mg/kg IV on Days 1, 8, 15, and 22 of Cycles 1 through 3 and then Days 1 and 15 of each 28-day cycle from Cycle 4 onward. Participants also self-administered parsaclisib at a dose of 20 mg QD for 8 weeks, followed by a dose of 2.5 mg QD thereafter. Study treatment was administered until progression of disease, withdrawal of consent, or unacceptable toxicity.
- Cohort 4: R/R MZL: Participants with R/R marginal zone lymphoma (MZL) received tafasitamab administered at 12 mg/kg IV on Days 1, 8, 15, and 22 of Cycles 1 through 3 and then Days 1 and 15 of each 28-day cycle from Cycle 4 onward. Participants also self-administered parsaclisib at a dose of 20 mg QD for 8 weeks, followed by a dose of 2.5 mg QD thereafter. Study treatment was administered until progression of disease, withdrawal of consent, or unacceptable toxicity.
- Cohort 5: R/R CLL/SLL: Participants with R/R chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) received tafasitamab administered at 12 mg/kg IV on Days 1, 8, 15, and 22 of Cycles 1 through 3 and then Days 1 and 15 of each 28-day cycle from Cycle 4 onward. Participants also self-administered parsaclisib at a dose of 20 mg QD for 8 weeks, followed by a dose of 2.5 mg QD thereafter. Study treatment was administered until progression of disease, withdrawal of consent, or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort 1: R/R DLBCL | Cohort 2: R/R MCL | Cohort 3: R/R FL | Cohort 4: R/R MZL | Cohort 5: R/R CLL/SLL
Started | 15 | 11 | 21 | 3 | 4
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 15 | 11 | 21 | 3 | 4
Not completed — Death | 9 | 7 | 4 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 1 | 0
Not completed — Sponsor Terminated Collection of Follow-up Data | 3 | 2 | 10 | 1 | 2
Not completed — Medical Decision Due to Worsening Clinical Condition | 1 | 0 | 0 | 0 | 0
Not completed — Transitioned to Rollover Protocol | 0 | 1 | 2 | 0 | 1
Not completed — Withdrawal per Principal Investigator; New Treatment | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: R/R DLBCL | Cohort 2: R/R MCL | Cohort 3: R/R FL | Cohort 4: R/R MZL | Cohort 5: R/R CLL/SLL | Total
Number analyzed (Participants) | 15 | 11 | 21 | 3 | 4 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (15.47) | 68.9 (15.06) | 66.8 (8.03) | 65.7 (17.21) | 70.3 (5.74) | 67.5 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 11 | 3 | 2 | 22
  Male | 10 | 10 | 10 | 0 | 2 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 1 | 0 | 7
  Not Hispanic or Latino | 13 | 6 | 16 | 2 | 2 | 39
  Unknown or Not Reported | 1 | 2 | 3 | 0 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 14 | 9 | 18 | 3 | 3 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3 | 0 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE )
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE is any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until 90 days after the last dose of study drug.
Time Frame: up to 1092 days
Population: Full Analysis Set: all participants who received at least 1 dose of tafasitamab or parsaclisib
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: R/R DLBCL | Cohort 2: R/R MCL | Cohort 3: R/R FL | Cohort 4: R/R MZL | Cohort 5: R/R CLL/SLL
Number analyzed (Participants) | 15 | 11 | 21 | 3 | 4
Participants | 15 | 11 | 21 | 3 | 4

2. Primary Outcome: Number of Participants With Any ≥Grade 3 TEAE
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. A TEAE is any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until 90 days after the last dose of study drug. The severity of AEs was assessed using CTCAE v5.0 Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to 1092 days
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: R/R DLBCL | Cohort 2: R/R MCL | Cohort 3: R/R FL | Cohort 4: R/R MZL | Cohort 5: R/R CLL/SLL
Number analyzed (Participants) | 15 | 11 | 21 | 3 | 4
Participants | 12 | 9 | 18 | 3 | 2

3. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as the occurrence of any protocol-defined toxicity up to and including Day 28 (Cycle 1/Day 28), except those with a clear alternative explanation.
Time Frame: up to 28 days
Population: Dose-limiting Toxicity Evaluable Population: all participants who received at least 3 of 4 doses of tafasitamab and 21 days of treatment with parsaclisib 20 mg QD during the first cycle (28 days) or experienced a DLT
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: R/R DLBCL | Cohort 2: R/R MCL | Cohort 3: R/R FL | Cohort 4: R/R MZL | Cohort 5: R/R CLL/SLL
Number analyzed (Participants) | 15 | 11 | 21 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Objective Response Rate Based on Investigator Assessment: Percentage of Participants With CR/CMR or PR/PMR According to Lugano Criteria for NHL and International Working Group for Chronic Lymphocytic Leukemia (iwCLL) Criteria for CLL
Description: Lugano complete response/complete metabolic response (CR/CMR): target nodes/masses of lymph nodes/extralymphatic sites (LNs/ELSs) regressed to ≤1.5 cm; no non-measured lesions; organ enlargement regressed to normal; no new lesions (NNLs); normal bone marrow. Lugano partial response/partial metabolic response (PR/PMR): LNs/ELSs, ≥50% decrease in the product of perpendicular diameters sum for multiple lesions; no/regressed non-measured lesions, no increase; organ enlargement; NNLs. iwCLL CR: no LNs ≥1.5 cm; spleen size <13 cm/liver size normal; no constitutional symptoms; normal circulating lymphocyte count (CLC); ≥100 × 10^9 platelets/L; hemoglobin ≥11 g/dL; normocellular, no CLL cells, no B-lymphoid nodules in marrow. iwCLL PR decrease of ≥50% in lymph nodes, liver and/or spleen, and CLC from baseline; constitutional symptoms; ≥100 × 10^9 platelets/L or increase of ≥50% over baseline in platelet count and hemoglobin; presence of CLL cells, or of B-lymphoid nodules, or not done.
Time Frame: up to 1002 days
Population: Full Analysis Set. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: R/R DLBCL | Cohort 2: R/R MCL | Cohort 3: R/R FL | Cohort 4: R/R MZL | Cohort 5: R/R CLL/SLL
Number analyzed (Participants) | 15 | 11 | 21 | 3 | 4
percentage of participants | 33.3 [11.8 to 61.6] | 81.8 [48.2 to 97.7] | 90.5 [69.6 to 98.8] | 33.3 [0.8 to 90.6] | 50.0 [6.8 to 93.2]

5. Secondary Outcome: Cmax of Tafasitamab When Given in Combination With Parsaclisib
Description: Cmax was defined as the maximum observed plasma or serum concentration of tafasitamab.
Time Frame: Cycle 1 Day 1; before tafasitamab infusion (predose); immediately after tafasitamab infusion; 1 hour and 4 hours post-infusion
Population: Pharmacokinetic (PK) Evaluable Population: all participants who received at least 1 dose of tafasitamab or parsaclisib and provided at least 1 postdose PK plasma sample. PK is not influenced by different oncology indications; thus, PK data were not analyzed by individual oncology cohorts.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Groups:
- All Cohorts: Participants with R/R DLBCL, R/R, MCL, R/R FL, R/R MZL, and CLL/SLL received tafasitamab administered at 12 mg/kg IV on Days 1, 8, 15, and 22 of Cycles 1 through 3 and then Days 1 and 15 of each 28-day cycle from Cycle 4 onward. Participants also self-administered parsaclisib at a dose of 20 mg QD for 8 weeks, followed by a dose of 2.5 mg QD thereafter. Study treatment was administered until progression of disease, withdrawal of consent, or unacceptable toxicity.
Arm/Group | All Cohorts
Number analyzed (Participants) | 53
milligrams per liter (mg/L) | 324.203 (112.746)

6. Secondary Outcome: Tmax of Tafasitamab When Given in Combination With Parsaclisib
Description: tmax was defined as the time to the maximum concentration of tafasitamab.
Time Frame: as for outcome 5
Population: PK Population. PK is not influenced by different oncology indications; thus, PK data were not analyzed by individual oncology cohorts.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | All Cohorts
Number analyzed (Participants) | 53
hours | 3.963 (1.591)

7. Secondary Outcome: AUClast of Tafasitamab When Given in Combination With Parsaclisib
Description: AUClast was defined as the area under the plasma concentration-time curve from time zero to the time of the last measurable concentration.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours x mg/L
Arm/Group | All Cohorts
Number analyzed (Participants) | 53
hours x mg/L | 31379.84 (12369.81)

8. Secondary Outcome: AUC0-inf of Tafasitamab When Given in Combination With Parsaclisib
Description: AUC0-inf was defined as the area under the plasma concentration-time curve from time zero to infinity (time that the drug is no longer present in the body).
Time Frame: as for outcome 5
Population: PK Population. Only participants with available data were analyzed. PK is not influenced by different oncology indications; thus, PK data were not analyzed by individual oncology cohorts.
Measure: Mean (Standard Deviation); unit: hours x mg/L
Arm/Group | All Cohorts
Number analyzed (Participants) | 51
hours x mg/L | 54825.21 (29363.32)

9. Secondary Outcome: Clast of Tafasitamab When Given in Combination With Parsaclisib
Description: AUC0-inf was defined as the last measurable plasma drug concentration.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | All Cohorts
Number analyzed (Participants) | 53
mg/L | 114.386 (56.789)

10. Secondary Outcome: t1/2 of Tafasitamab When Given in Combination With Parsaclisib
Description: t1/2 was defined as the drug's elimination half-life, which is the time it takes for the concentration of a drug in the body to decrease by 50%.
Time Frame: as for outcome 5
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | All Cohorts
Number analyzed (Participants) | 51
hours | 121.702 (49.506)

11. Secondary Outcome: CL of Tafasitamab When Given in Combination With Parsaclisib
Description: CL was defined as the apparent total body clearance of drug from plasma.
Time Frame: as for outcome 5
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | All Cohorts
Number analyzed (Participants) | 51
liter per hour | 0.021 (0.015)

12. Secondary Outcome: VZ of Tafasitamab When Given in Combination With Parsaclisib
Description: Vz was defined as the volume of distribution.
Time Frame: as for outcome 5
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | All Cohorts
Number analyzed (Participants) | 51
liters | 3.254 (1.694)

ADVERSE EVENTS:
Time Frame: up to 1092 days
Description: Adverse events have been reported for the Full Analysis Set, comprised of all participants who received at least 1 dose of tafasitamab or parsaclisib.
Arm/Group | Cohort 1: R/R DLBCL | Cohort 2: R/R MCL | Cohort 3: R/R FL | Cohort 4: R/R MZL | Cohort 5: R/R CLL/SLL
All-Cause Mortality (participants affected / at risk) | 9/15 | 7/11 | 4/21 | 0/3 | 1/4
Serious Adverse Events (participants affected / at risk) | 6/15 | 7/11 | 12/21 | 2/3 | 3/4
Other Adverse Events (participants affected / at risk) | 15/15 | 11/11 | 21/21 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: R/R DLBCL (N=15) | Cohort 2: R/R MCL (N=11) | Cohort 3: R/R FL (N=21) | Cohort 4: R/R MZL (N=3) | Cohort 5: R/R CLL/SLL (N=4)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (7) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: R/R DLBCL (N=15) | Cohort 2: R/R MCL (N=11) | Cohort 3: R/R FL (N=21) | Cohort 4: R/R MZL (N=3) | Cohort 5: R/R CLL/SLL (N=4)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (5) | 2 (2) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 5 (5) | 3 (6) | 6 (7) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (4) | 1 (2) | 8 (10) | 1 (1) | 2 (2)
Campylobacter colitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (6) | 2 (2) | 0 (0) | 3 (4)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (3) | 3 (4) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 2 (2) | 11 (15) | 2 (3) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Dysgraphia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (4)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (9) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 7 (12) | 6 (11) | 11 (19) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
POEMS syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic bone injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (5) | 3 (3) | 6 (9) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 7 (8) | 3 (4) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (4) | 2 (2) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Xerosis (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The sponsor chose to terminate the study early due to the strategic business decision to discontinue the evaluation of parsaclisib in clinical studies. Participants who continued to receive clinical benefit (in the opinion of the investigator) had the option to transition to a rollover study for continued supply of parsaclisib in combination with tafasitamab (including supply of tafasitamab to those who remained on tafasitamab alone).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT04809467/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT04809467/SAP_001.pdf